CLINICAL TRIAL: NCT02364284
Title: Reporting Patterns and Results of Initial Antibiotic Treatment in Patients With Complicated Urinary Tract Infection,Complicated Intra-abdominal Infection and Nosocomial Pneumonia Including Ventilator-associated Pneumonia.
Brief Title: Reporting Patterns and Results of Initial Antibiotic Treatment in Patients With cUTI, cIAI,NP Including VAP
Acronym: RECOMMEND
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: D4280R00005
Record Dates: First submitted 2015-02-06; First posted 2015-02-18 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Urinary Tract Infection (cUTI); Intra-abdominal Infection (cIAI) and; Nosocomial Pneumonia (NP)
MeSH Terms: conditions — Urinary Tract Infections; Intraabdominal Infections; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Urinary Tract Infection (cUTI): Patients ≥18 years with diagnosis of urinary tract infection.
- Intra Abdominal Infection(cIAI): Patients ≥ 18 years with diagnosis of Intra Abdominal Infection
- Nosocomial Pneumonia (NP): Patients ≥ 18 years with diagnosis of Hospital acquired pneumonia

SUMMARY:
Reporting patterns and results of initial antibiotic treatment in patients with complicated urinary tract infection (cUTI), complicated intra-abdominal infection (cIAI) and nosocomial pneumonia (NP) including ventilator-associated pneumonia (VAP) - RECOMMEND Study

DETAILED DESCRIPTION:
This will be an observational, historical cohort study from medical chart review of adult hospitalized patients for each of the three conditions of interest (complicated urinary tract infection (cUTI), complicated intra-abdominal infection (cIAI) and nosocomial pneumonia (NP) including ventilator-associated pneumonia (VAP)). For this study, the proposed patient selection period extends for 12 months, from July 1, 2013 to June 30, 2014. Patients selected during this period will be followed from diagnosis (i.e., diagnosis of cUTI, cIAI or NP) until symptom resolution, discharge or 30-days post discharge [based on data availability to assess readmission and outpatient visits], death while hospitalized, loss to follow-up or the end of study period if not yet discharged from index hospitalization [December 31, 2014]).

ELIGIBILITY:
Inclusion Criteria:

ICF to be obtained (refer slides 26-30) Adult (≥18 years) patients Patients with a diagnosis of at least one of the three conditions hospitalised during the period July 1, 2013 to June 30, 2014 Hospital acquired or healthcare associated cUTI Hospital acquired or healthcare associated cIAI NP including VAP

Exclusion Criteria:

The patient participated in a clinical trial during the patient selection period (01-Jul-2013 to 30-Jun-2014) or during the follow-up period* For patients diagnosed with cUTI: The patient has a diagnosis of hospital acquired or healthcare associated cUTI with concomitant presence of Fungal UTI with colony count > 10^3/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) patients. Hospitalized patients with a diagnosis of at least one of the following three conditions during the period July 1, 2013 to June 30, 2014 should be included in this study.
  Hospital acquired or healthcare associated cUTI Hospital acquired or healthcare associated cIAI NP including VAP
Sampling Method: Non-Probability Sample
Enrollment: 1322 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To describe antibiotic management and document treatment outcome among hospitalized patients with hospital acquired or healthcare associated cUTI, cIAI and NP | 12 months
  Evaluate failure or success of the initial antibiotic treatment following cUTI, cIAI and NP diagnosis. Initial antibiotic therapy is defined as all antibiotic agents received during the 48 hours post initiation of antibiotic therapy - The primary outcome measure will be assessed from the antibiotic initiation date until end of follow-up defined by in-hospital with symptom resolution, in-hospital without symptom resolution, discharged to home, discharged to other health care facility, readmission within 30 days for same infection, readmission within 30 days post discharge with other diagnosis, death during hospital stay, death post discharge within 30 days.

SECONDARY OUTCOMES:
To identify potential risk factors related to outcomes of initial antibiotic treatment of hospitalized patients with hospital acquired or healthcare associated cUTI, cIAI and NP | 12 months
  Assess risk factors related to the primary outcome measure. Covariates considered in the risk assessment will include: site characteristics, patient characteristics, secondary infections, prior medical history and comorbidity burden, hospitalization characteristics, pathogen characteristics, co-medications - The listed covariates will be assessed at baseline (i.e., at index hospitalization date), during the hospital stay and the 30-day period post discharge date.
To describe healthcare utilization and costs associated with hospital acquired or healthcare associated cUTI, cIAI and NP initial antibiotic treatment outcome | 12 months
  Assess health care utilization among patients with cUTI, cIAI and NP. Variables assessed to address this will include - hospital length of stay, ICU length of stay, number of surgical procedures, number of outpatient visits, days on antibiotic therapy, number of readmission during follow-up - The listed measures will be assessed during the hospital stay and during the 30-day period post discharge date.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Fedou, Principal Investigator — CHU de Limoges - Hôpital Dupuytren
Locations (27):
- Brazil (3):
  - Research Site, Belo Horizonte
  - Research Site, Campinas
  - Research Site, Porto Alegre
- France (6):
  - Research Site, Argenteuil
  - Research Site, Bordeaux
  - Research Site, Créteil
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Nantes
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Italy (5):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Monza
  - Research Site, Roma
  - Research Site, Vicenza
- Russia (4):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Sestroretsk, Saint Petersburg
- Spain (5):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Oviedo
  - Research Site, Seville
  - Research Site, Terrassa

REFERENCES:
- [Derived] Ryan K, Karve S, Peeters P, Baelen E, Potter D, Rojas-Farreras S, Pascual E, Rodriguez-Bano J. The impact of initial antibiotic treatment failure: Real-world insights in healthcare-associated or nosocomial pneumonia. J Infect. 2018 Jul;77(1):9-17. doi: 10.1016/j.jinf.2018.04.002. Epub 2018 May 6. PMID 29742471
- [Derived] Karve S, Ryan K, Peeters P, Baelen E, Rojas-Farreras S, Potter D, Rodriguez-Bano J. The impact of initial antibiotic treatment failure: Real-world insights in patients with complicated urinary tract infection. J Infect. 2018 Feb;76(2):121-131. doi: 10.1016/j.jinf.2017.11.001. Epub 2017 Nov 8. PMID 29128389
- See also: D4280R00005_RECOMMEND_CSR_Synopsis_17Nov2016(redacted)_final — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2972&filename=D4280R00005_RECOMMEND_CSR_Synopsis_17Nov2016(redacted)_final.pdf